CLINICAL TRIAL: NCT05203120
Title: A National Phase II Study of Proton Therapy in Hepatocellular Carcinoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Herlev Hospital (Other); Rigshospitalet, Denmark (Other); Odense University Hospital (Other); University of Leeds (Other); Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCPT HCC
Record Dates: First submitted 2021-12-13; First posted 2022-01-24 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Proton Therapy

STUDY DESIGN:
Intervention Model Description: National phase II non-randomized single-arm study of proton therapy in patients with hepatocellular carcinoma.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Proton Arm (Experimental): All patients in the study will receive proton therapy with 67.5 Gray/15 fractions(fx) /5fx per week .
  Interventions: Radiation: Proton therapy

INTERVENTIONS:
Radiation: Proton therapy — All patients will receive proton therapy 67.5Gy/15fx

SUMMARY:
350 new cases of hepatocellular carcinoma (HCC) are diagnosed in Denmark each year, but the overall prognosis is poor with a 1-year survival rate of less than 40% and a 5-year survival rate of 10% for the entire patient group.

This national phase II non-randomized single-arm study of proton therapy in HCC is conducted with the aim to offer a safe and efficient radiation treatment to fragile patients with reduced dose to the normal liver compared to conventional photon-based radiotherapy.

DETAILED DESCRIPTION:
Each year, approximately 350 new cases of hepatocellular carcinoma (HCC) are diagnosed in Denmark, but the overall prognosis is poor with a 1-year survival rate of less than 40% and a 5-year survival rate of 10% for the entire patient group.

This national phase II non-randomized single-arm study of proton therapy in HCC is conducted with the aim to offer a safe and efficient radiation treatment to fragile patients with reduced dose to the normal liver compared to conventional photon-based radiotherapy. The study aims to offer curative treatment to a larger group of patients and thus better prognosis for these patients.

The study will include 50 patients enrolled within 3 years. Patients cannot be guaranteed any direct personal benefits of participating in the trial. Participating in the study can help with new knowledge that can benefit future patients with similar illness.

The treatment will be given at the Danish Center for Particle Therapy. During radiotherapy, additional CT scans will be performed weekly as part of quality assurance until it can be documented that there is no such need.

Participation in the study will also mean additional examinations and questionnaires at the start of treatment, below treatment and at follow-up.

All patients will be asked to supply blood samples to analyze for circulating tumor DNA.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCC based on classical radiologic findings as defined by the American Association for the Study of Liver Diseases (AASLD) criteria or verified by biopsy
* No extra-hepatic disease
* Deemed ineligible for resection or Radiofrequency Ablation (RFA), or the patients should refuse RFA or surgery
* Age ≥ 18 years
* Performance status ≤ 2
* Total diameter of tumor(s) ≤ 12 cm and a maximum of 3 tumors
* Adequate liver function as measured by Child-Pugh score (Child-Pugh score ≤ 8), or absence of cirrhosis
* Has recovered adequately from toxicity and/or complications from any previous local interventions
* Patients with past or ongoing hepatitis C infection are allowed, but treatment for hepatitis C must have been completed one month before study entry
* Patients with hepatitis B infection is allowed if antiviral therapy have been given for at least 4 weeks and Hepatitis B Virus (HBV) viral load is less than 100 IU/ml. The active therapy must continue throughout the radiation therapy. Patients who are Total hepatitis B core antibody (anti-HBc)(+), negative for Hepatitis B surface antigen (HbsAg) and negative or positive for Hepatitis B surface antibody (anti-HBs) with a HBV viral load under 100 IU/mL do not require HBV anti-viral prophylaxis
* Adequate organ function

  * hematological: hemoglobin ≥ 6 mmol/l, absolute neutrophil count (ANC) ≥ 1,5 x 109/L, platelets ≥ 50 x 109/L
  * hepatic: bilirubin ≤ 1.5 x ULN, alanin-aminotransferase (ALAT) ≤ 1.5 x ULN
  * renal: creatinine ≤ 1.5 x ULN
* Ability to adhere to procedures for study and follow-up
* Signed informed consent to participate
* Final decisions on inclusion and treatment with proton therapy are at the discretion of the investigator

Exclusion Criteria:

* Previous x-ray-based radiotherapy in the liver
* Child Pugh score >8
* Tumor less than 1 cm from any critical organs at risk (OAR) (duodenum, kidney, stomach, intestines).
* Previous Selective internal radiation therapy (SIRT)
* Episode of hepatic encephalopathy within the last 6 months
* Uncontrolled ascites with need for drainage > 1 per month
* Episode of bleeding esophageal varices within the past month. If active bleeding from esophageal varices has occurred, a gastroscopy should be performed 4 weeks after the bleeding episode to ensure maximum grade 1 varices.
* Patients with metal implants where beam entrance through the metal implants cannot be avoided (not applicable for fiducial markers implanted for radiotherapy use)
* Patients for whom it is not possible to produce a robust treatment plan following the technical guidelines (Appendix A)
* Patients for whom it is not possible to implant fiducial markers e.g. due to insufficient coagulation of the blood.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Number of deaths of any cause | 4 months after start of radiotherapy
  Death of any cause
Number of participants with Radiation-induced liver disease (RILD) | 4 months after start of radiotherapy
  Worsening of the Child- Pugh score ≥2 or alanin-aminotransferase (ALAT) ≥5 upper normal limit (ULN)

SECONDARY OUTCOMES:
Number of participants with RILD within 6 months of start of radiotherapy | 6 months after start of radiotherapy
  Worsening of the Child- Pugh score ≥2 or ALAT ≥5 ULN
Acute toxicity | 4 months after start of radiotherapy
  Number of participants with Acute radiation-related toxicity grade 3 or higher measured by CTCAE v5.0
Late toxicity | from 4 months until 60 months after start of radiotherapy
  Number of participants with Late radiation-related toxicity grade 3 or higher measured by CTCAE v5.0
Radiation-induced hospitalization | within 4 months after start of radiotherapy
  Number of days spend in the hospital due to radiotherapy toxicity
Health-related Quality of Life C30 | Until 60 months after start of radiotherapy
  Health-related Quality of life measured by the EORTC QoL questionnaires C30
Quality of Life HCC-18 | Until 60 months after start of radiotherapy
  Health-related Quality of life measured by the EORTC QoL questionnaires HCC18
Local control | 3 years after start of radiotherapy
  1- and 3-year local control
Progression-free survival | 3 years after start of radiotherapy
  1- and 3-year progression-free survival
Overall survival | 3 years after start of radiotherapy
  1- and 3-year overall survival
Pattern of failure | Until 5 years after start of radiotherapy
  Pattern of failure will be reported as number of patients with in-field failures in the clinical target volumen (CTV), in-field failures in the planning target volume (PTV), and out-of-field failures.
Technical feasibility | up to 5 years
  the proportion of patients where it was possible to adhere to the guidelines of CTV dose coverage and tolerable normal tissue dose
Reduction in mean liver dose | up to 5 years
  calculated on a per patient basis, and median (and inter-quartile ranged) will be reported for the study population.

CONTACTS AND LOCATIONS:
Overall Officials: Britta Weber, MD PhD, Principal Investigator — Danish Center of Particle Therapy
Locations (3):
- Denmark (3):
  - Herlev Hospital, Herlev, Capital Region
  - Aarhus University Hospital, Aarhus, Central Jutland
  - Odense University Hospital, Odense, Syd

IPD SHARING:
Plan to Share IPD: No